CLINICAL TRIAL: NCT03834168
Title: The Diurnal Rhythm in Natriuretic Peptide Levels and Relationship With Nocturnal Blood Pressure
Brief Title: The Diurnal Rhythm in Natriuretic Peptide Levels
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Pankaj Arora, MD, Assistant Professor, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IRB-300002114
Record Dates: First submitted 2019-02-06; First posted 2019-02-07 (Actual); Results first posted 2021-08-31 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2024-01

CONDITIONS: Natriuretic Peptides; Obesity; Nocturnal Blood Pressure
Keywords: Diurnal Rhythm; Race
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study Individuals (Other): Healthy self-identified African-American and white male participants will be screened. Study consent will be obtained, medical history and physical examination administered, and study eligibility determined based on the inclusion and exclusion criteria. Eligible subjects will meet a bio-nutritionist who will explain the 5 days of standardized diet at the screening visit and will review instructions for complying with the diet. If the subject agrees to adhere to the study diet, they will then be enrolled in the study (stratified by race).
  Interventions: Other: standardized Study Diet

INTERVENTIONS:
Other: standardized Study Diet — Standardized diet consisted with eucaloric meals with 4.5 gm of sodium per day for 5 days.

SUMMARY:
The purpose of the study to assess the diurnal rhythm in natriuretic peptide levels and its temporal relationship with nocturnal blood pressure in obese and African-American individuals as compared with lean and white individuals.

DETAILED DESCRIPTION:
Obese and African-American individuals are at greater risk for cardiovascular morbidity and mortality than lean and white individuals. One of the key reasons for this health disparity is a higher risk of hypertension among obese and African-American individuals. The reasons for why these disparities develop are not well understood.

Natriuretic peptides are hormones produced by the heart and have a wide range of favorable cardiovascular effects such as natriuresis (sodium excretion), vasodilation, and direct inhibition of the renin-angiotensin-aldosterone system. Human studies showed the existence of 24-hour (diurnal) variations in the circulating natriuretic peptide levels.

Prior work from the investigators and others demonstrated that individuals with genetically-determined lower circulating natriuretic peptides levels have higher blood pressure and greater risk of hypertension. Further, the investigators have shown that obesity and African-American race are associated with lower natriuretic peptide levels, suggesting that relatively low natriuretic peptide levels may be a biologic determinant contributing to health disparities.

Obese and African-American individuals have a greater prevalence of nocturnal hypertension [nighttime blood pressure >120/80 mmHg], which is an independent risk factor for cardiovascular events. The underlying reasons for 24-hour variations in blood pressure are unknown.

The investigators hypothesize that loss of the natural 24-hour rhythm of natriuretic peptide levels plays a role in the development of nocturnal hypertension in obese and African-American individuals. The aims of this study are:

1. to examine whether there is a presence of a 24-hour rhythm in natriuretic peptide levels among normotensive obese and African-American individuals and whether there is a difference in the rhythmicity of natriuretic peptide levels between obese and lean as well as in African-Americans and whites;
2. to examine whether there is an existence of a relationship between 24-hour variability of natriuretic peptide levels and 24-hour patterns of blood pressure and whether this relationship of rhythmicity of natriuretic peptide levels and nocturnal blood pressure differed in obese and lean individuals and by race.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 40 years
* Blood pressure less than 140/90
* Body Mass Index between 18.5 to 25 kg/m2 (lean) or 30 to 45 kg/m2 (obese)
* Self identified African-American or white individuals
* Willingness to comply with the study diet
* Provide informed consent

Exclusion Criteria:

* History of hypertension
* History of cardiovascular, renal, or liver disease
* Diabetes or use of glucose-lowering medications
* Use of vasoactive or diuretic medications
* Atrial fibrillation
* Anemia (Hematocrit <41%)
* Abnormal serum sodium or potassium
* Abnormal liver function tests (>3x upper limit of normal)
* Current smokers
* Regular users of non-steroid anti-inflammatory medications

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-02-29 (Actual); Study Completion 2021-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pankaj Arora, MD, Principal Investigator — University of Alabama at Birmingham; Orlando M Gutierrez, MMSc, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Goetze JP, Jorgensen HL, Sennels HP, Fahrenkrug J. Diurnal plasma concentrations of natriuretic propeptides in healthy young males. Clin Chem. 2012 Apr;58(4):789-92. doi: 10.1373/clinchem.2011.178921. Epub 2012 Jan 26. No abstract available. PMID 22282468
- [Background] Arora P, Reingold J, Baggish A, Guanaga DP, Wu C, Ghorbani A, Song Y, Chen-Tournaux A, Khan AM, Tainsh LT, Buys ES, Williams JS, Heublein DM, Burnett JC, Semigran MJ, Bloch KD, Scherrer-Crosbie M, Newton-Cheh C, Kaplan LM, Wang TJ. Weight loss, saline loading, and the natriuretic peptide system. J Am Heart Assoc. 2015 Jan 16;4(1):e001265. doi: 10.1161/JAHA.114.001265. PMID 25595796
- [Background] Bajaj NS, Gutierrez OM, Arora G, Judd SE, Patel N, Bennett A, Prabhu SD, Howard G, Howard VJ, Cushman M, Arora P. Racial Differences in Plasma Levels of N-Terminal Pro-B-Type Natriuretic Peptide and Outcomes: The Reasons for Geographic and Racial Differences in Stroke (REGARDS) Study. JAMA Cardiol. 2018 Jan 1;3(1):11-17. doi: 10.1001/jamacardio.2017.4207. PMID 29167879
- [Background] Arora P, Wu C, Hamid T, Arora G, Agha O, Allen K, Tainsh RET, Hu D, Ryan RA, Domian IJ, Buys ES, Bloch DB, Prabhu SD, Bloch KD, Newton-Cheh C, Wang TJ. Acute Metabolic Influences on the Natriuretic Peptide System in Humans. J Am Coll Cardiol. 2016 Feb 23;67(7):804-812. doi: 10.1016/j.jacc.2015.11.049. PMID 26892417
- [Result] Parcha V, Patel N, Gutierrez OM, Li P, Gamble KL, Musunuru K, Margulies KB, Cappola TP, Wang TJ, Arora G, Arora P. Chronobiology of Natriuretic Peptides and Blood Pressure in Lean and Obese Individuals. J Am Coll Cardiol. 2021 May 11;77(18):2291-2303. doi: 10.1016/j.jacc.2021.03.291. PMID 33958126

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 42 participants agreed to participate in the study following the completion of the informed consent process and were assigned to each Arm/group. We had one study dropout and one participant was not able to complete the protocol. A total of 40 participants completed the study.
Groups:
- Lean: Healthy self-identified African-American and white male lean participants will be screened. Study consent will be obtained, medical history and physical examination administered, and study eligibility determined based on the inclusion and exclusion criteria. Eligible subjects will meet a bio-nutritionist who will explain the 5 days of standardized diet at the screening visit and will review instructions for complying with the diet. If the subject agrees to adhere to the study diet, they will then be enrolled in the study (stratified by race).
  standardized Study Diet: Standardized diet consisted with eucaloric meals with 4.5 gm of sodium per day for 5 days.
- Obese: Healthy self-identified African-American and white male obese participants will be screened. Study consent will be obtained, medical history and physical examination administered, and study eligibility determined based on the inclusion and exclusion criteria. Eligible subjects will meet a bio-nutritionist who will explain the 5 days of standardized diet at the screening visit and will review instructions for complying with the diet. If the subject agrees to adhere to the study diet, they will then be enrolled in the study (stratified by race).
  standardized Study Diet: Standardized diet consisted with eucaloric meals with 4.5 gm of sodium per day for 5 days.
Period: Overall Study
Arm/Group | Lean | Obese
Started (42 participants started the study; 19 Lean and 23 Obese) | 19 | 23
Total Participant Screened for the Purpose of Eligibility (52 Participants were screened for the eligibilty) | 22 | 30
Ineligible Participants (10 participants determined ineligible by screening labs) | 3 | 7
Unable to Complete the Protocol | 0 | 1
Study Dropouts | 1 | 0
Participants Received 5 Days of Standardized Meals (42 participants received 5 days of standardized meals to control the salt intake) | 19 | 23
Participants Returned for the 24-h Inpatient Protocol (41 participants returned for the 24-h inpatient protocol) | 18 | 23
Completed (40 participants completed the study; 18 Lean and 22 Obese) | 18 | 22
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Lean: Healthy self-identified African-American and white lean participants will be screened. Study consent will be obtained, medical history and physical examination administered, and study eligibility determined based on the inclusion and exclusion criteria. Eligible subjects will meet a bio-nutritionist who will explain the 5 days of standardized diet at the screening visit and will review instructions for complying with the diet. If the subject agrees to adhere to the study diet, they will then be enrolled in the study (stratified by race).
  standardized Study Diet: Standardized diet consisted with eucaloric meals with 4.5 gm of sodium per day for 5 days.
- Obese: Healthy self-identified African-American and white obese participants will be screened. Study consent will be obtained, medical history and physical examination administered, and study eligibility determined based on the inclusion and exclusion criteria. Eligible subjects will meet a bio-nutritionist who will explain the 5 days of standardized diet at the screening visit and will review instructions for complying with the diet. If the subject agrees to adhere to the study diet, they will then be enrolled in the study (stratified by race).
  standardized Study Diet: Standardized diet consisted with eucaloric meals with 4.5 gm of sodium per day for 5 days.
- Total: Total of all reporting groups
Arm/Group | Lean | Obese | Total
Number analyzed (Participants) | 18 | 22 | 40
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 30.5 [24.0 to 32.0] | 33.0 [26.0 to 37.0] | 31.0 [26.0 to 35.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 12 | 20
  Male | 10 | 10 | 20
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 10 | 16 | 26
  White | 0 | 0 | 0
  More than one race | 8 | 6 | 14
  Unknown or Not Reported | 0 | 0 | 0
Body Mass Index [Median (Inter-Quartile Range); unit: kg/m^2] | 24.3 [21.9 to 25.0] | 32.2 [30.7 to 36.0] | 29.6 [24.4 to 32.9]
Hip circumference [Median (Inter-Quartile Range); unit: cm] | 97.3 [93.8 to 101.0] | 111.4 [106.1 to 118.7] | 106.1 [96.1 to 114.8]
Waist circumference [Median (Inter-Quartile Range); unit: cm] | 76.9 [73.5 to 85.7] | 103.6 [99.8 to 111.8] | 97.6 [78.3 to 105.4]
Systolic Blood Pressure [Median (Inter-Quartile Range); unit: mmHg] | 110.7 [102.0 to 122.7] | 116.5 [108.3 to 126.0] | 116.2 [106.0 to 123.0]
Diastolic Blood Pressure [Median (Inter-Quartile Range); unit: mmHg] | 69.5 [64.3 to 76.0] | 73.7 [67.7 to 80.0] | 71.0 [65.3 to 78.2]
Heart rate [Median (Inter-Quartile Range); unit: beats/min] | 76.5 [66.0 to 80.0] | 77.0 [71.0 to 80.0] | 77.0 [69.0 to 80.0]
Fasting Glucose [Median (Inter-Quartile Range); unit: mg/dL] | 85.0 [79.0 to 96.0] | 91.5 [82.0 to 100.0] | 87.5 [81.0 to 97.0]
Renal Function [Median (Inter-Quartile Range); unit: mg/dL]
  Blood Urea Nitrogen (BUN) | 12.0 [11.0 to 13.0] | 12.0 [10.0 to 14.0] | 12 [10.5 to 14.0]
  Serum Creatinine | 0.9 [0.8 to 0.9] | 0.9 [0.8 to 1.0] | 0.9 [0.8 to 0.9]
Serum Electrolytes [Median (Inter-Quartile Range); unit: mEq/L]
  Sodium, mEq/L | 137.5 [137.0 to 139.0] | 138.0 [136.0 to 138.0] | 138.0 [136.5 to 138.5]
  Potassium, mEq/L | 4.2 [3.9 to 4.3] | 4.2 [4.0 to 4.3] | 4.2 [3.9 to 4.3]
  Chloride, mEq/L | 102.5 [102.0 to 104.0] | 103.5 [102.0 to 105.0] | 103.0 [102.0 to 104.0]
  Bicarbonate, mEq/L | 26.0 [25.0 to 28.0] | 26.0 [25.0 to 27.0] | 26.0 [25.0 to 27.0]
Serum Calcium [Median (Inter-Quartile Range); unit: mg/dL] | 9.6 [9.3 to 9.7] | 9.6 [9.2 to 9.8] | 9.6 [9.3 to 9.7]
Liver Function [Median (Inter-Quartile Range); unit: mg/dL]
  Total bilirubin | 0.5 [0.4 to 0.8] | 0.5 [0.4 to 0.7] | 0.5 [0.4 to 0.8]
  Alanine transaminase (ALT) | 13.5 [11.0 to 16.0] | 17.0 [12.0 to 27.0] | 14.0 [12.0 to 20.0]
  Aspartate transaminase (AST) | 17.0 [14.0 to 20.0] | 17.0 [14.0 to 23.0] | 17.0 [14.0 to 20.0]
  Gamma-glutamyl transferase (GGT) | 16.0 [12.0 to 24.0] | 22.5 [15.0 to 27.0] | 20.0 [12.5 to 25.5]
Hematological Parameters [Median (Inter-Quartile Range); unit: cells*10,000/mm^3]
  WBC, * 10,000/mm3 | 5.3 [4.3 to 6.7] | 5.5 [4.6 to 6.1] | 5.4 [4.4 to 6.3]
  RBC, * 1,000,000/mm3 | 4.7 [4.1 to 5.0] | 4.7 [4.1 to 5.0] | 4.7 [4.1 to 5.0]
  Platelet, * 100,000/mm3 | 217.7 [192.8 to 274.9] | 248.7 [223.6 to 268.2] | 243.4 [202.2 to 271.6]
Hemoglobin [Median (Inter-Quartile Range); unit: g/dL] | 14.0 [13.1 to 14.9] | 14.2 [13.2 to 14.8] | 14.2 [13.2 to 14.8]
Hematocrit [Median (Inter-Quartile Range); unit: %] | 40.5 [37.0 to 43.0] | 41.0 [38.0 to 43.0] | 41.0 [37.5 to 43.0]
Mean Corpuscular Volume (MCV) [Median (Inter-Quartile Range); unit: fl] | 87.5 [84.0 to 90.0] | 89.0 [86.0 to 92.0] | 88.0 [86.0 to 91.0]
Mean Corpuscular Hemoglobin (MCH) [Median (Inter-Quartile Range); unit: pg] | 30.0 [29.0 to 31.0] | 31.0 [29.0 to 32.0] | 30.0 [29.0 to 31.0]
Mean Corpuscular Hemoglobin Concentration (MCHC) [Median (Inter-Quartile Range); unit: g/dL] | 34.0 [33.0 to 34.0] | 34.0 [33.0 to 35.0] | 34.0 [33.0 to 34.5]
Red Cell Distribution Width (RDW) [Median (Inter-Quartile Range); unit: %] | 13.5 [13.1 to 13.9] | 13.3 [12.8 to 14.5] | 13.5 [12.8 to 14.0]
Mean Platelet Volume (MPV) [Median (Inter-Quartile Range); unit: fL] | 9.0 [8.0 to 9.0] | 8.0 [8.0 to 9.0] | 9.0 [8.0 to 9.0]

OUTCOME MEASURES:

1. Primary Outcome: Plasma MRproANP
Description: Assess the diurnal rhythm in circulating MRproANP levels among obese individuals and compared it with lean individuals
Time Frame: About 24 hours on the in-patient study visit day after consuming study meals for 5 days
Measure: Median (Inter-Quartile Range); unit: pmol/l
Arm/Group | Lean | Obese
Number analyzed (Participants) | 18 | 22
pmol/l | 17.92 [12.94 to 25.21] | 15.51 [10.61 to 22.02]
Statistical Analysis 1: Comparison: Lean; Test type: Other; p = 0.003, Regression (Cosinor Fit)
Statistical Analysis 2: Comparison: Lean vs Obese; Test type: Superiority; p < 0.001, Regression, Linear

2. Secondary Outcome: Acrophase Difference in Hours Between the MR-proANP and Systolic BP Rhythm
Description: Assess relationship between 24-hour variability of MRproANP levels and 24-hour patterns of blood pressure and whether this relationship of rhythmicity of MRproANP levels and nocturnal blood pressure differed in obese and lean individuals and by race
Time Frame: About 24 hours on the in-patient study visit day after consuming study meals for 5 days
Measure: Mean (Standard Error); unit: Hours
Arm/Group | Lean | Obese
Number analyzed (Participants) | 18 | 22
Hours | -0.7 (0.03) | -4.9 (0.05)

3. Other Pre Specified Outcome: Plasma MRproANP
Description: Assess the diurnal rhythm in circulating MRproANP levels among African-American individuals and compared it with white individuals
Time Frame: About 24 hours on the in-patient study visit day after consuming study meals for 5 days
Population: The race-specific analysis was not done for this study
Arm/Group | Lean | Obese
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 month
Arm/Group | Lean | Obese
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/22
Other Adverse Events (participants affected / at risk) | 0/18 | 0/22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-01-20): https://cdn.clinicaltrials.gov/large-docs/68/NCT03834168/Prot_SAP_000.pdf
  • Informed Consent Form (2021-01-20): https://cdn.clinicaltrials.gov/large-docs/68/NCT03834168/ICF_001.pdf